CLINICAL TRIAL: NCT03895866
Title: Clinical Study on the Relationship Between Persistent Cervical HPV Infection With Clearance and Vaginal Microbial Community
Brief Title: Persistent Cervical HPV Infection With Clearance and Vaginal Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, shuwang, Associate Professor, Peking Union Medical College Hospital
Other Study IDs: HPV clearance
Record Dates: First submitted 2019-02-04; First posted 2019-03-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: HPV-Related Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: High-risk HPV persistent infection more than half a year and reversion
  Interventions: Other: The participants were assigned to different groups according to the results of HPV detection.
- Group B: High-risk HPV non-infection
  Interventions: Other: The participants were assigned to different groups according to the results of HPV detection.

INTERVENTIONS:
Other: The participants were assigned to different groups according to the results of HPV detection. — The participants were assigned to different groups according to the results of HPV detection

SUMMARY:
Since other genital infections enhance HIV susceptibility by inducing inflammation, the investigators study the relationship between the vaginal microbiota composition and the persistence infection and clearance of HPV infection.

DETAILED DESCRIPTION:
Persistent infection with oncogenic Human Papillomavirus (HPV) is necessary but not sufficient for the development of cervical cancer. Additional factors correlated with HPV persistence include immunodeficiency caused by HIV, smoking, use of oral contraceptives and, more recently reported, vaginal dysbiosis. In a state of dysbiosis, there is a marked reduction of Lactobacillus and a high diversity of bacteria, with increased abundance of anaerobic bacterial species. High-risk HPV cervical infections are common in young, sexually active women. Most of these infections are transient and do not cause clinical symptoms. After 12-30 months of HPV infection, 70-90% of patients can be cleared naturally, but there are still a small number of patients with high-risk HPV infection can not be eliminated by itself and continue to infect, and can develop into cervical intraepithelial neoplasia, eventually progressing to invasive cervical cancer. Persistent infection of high-risk HPV is a necessary condition for the occurrence of cervical cancer and precancerous lesions. Early blocking of persistent infection of high-risk HPV and timely treatment of cervical precancerous lesions are of great significance in preventing the occurrence of cervical cancer. This project intends to study the relationship between vaginal microbial composition and persistent HPV infection, and determine the related strains and their molecular mechanisms, so as to provide new ideas and basis for its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Those are aged 20 to 45 years old, have had vaginal intercourse more than 3 years, and aren't in menstrual, pregnancy or puerperium period.

Exclusion Criteria:

* Those have no vaginal intercourse, and can't cooperate the examiner. Women who are HIV or hepatitis B/C positive, have autoimmune disorders and systemic disease (like diabetes mellitus, hormone treatment diseases, severe liver and kidney dysfunction), or have severe mental illness and malignant tumors are also excluded. At the same time, all the participants should meet the following requirements: no vagina douching within last 2 days, no vaginal intercourse within last 3 days, no systemic application of antifungal agents or antibiotics or pessaries within last 14 days of sampling.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants sample was referred to the paper already published.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-02-11 (Estimated); Study Completion 2020-02-11 (Estimated)

PRIMARY OUTCOMES:
The relationship between diversity of vaginal microbiota and HR-HPV persistent infection | 12 months
  The persistent specific vaginal organism in HPV persistent infection women

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China